CLINICAL TRIAL: NCT00990275
Title: Alcohol Exposure and Airway Hyperresponsiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0268-07-FB; 1F32AA017024-01 (NIH)
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-alcohol change in airway hyperresponsiveness. (Experimental): Participants will ingest 3 ounces of vodka mixed with fruit juice within 30 min. Then provocative concentration causing a 20% fall in forced expiratory volume in 1 s (PC20FEV1) will be measured. A one-half concentration difference in the PC20FEV1 will be considered a statistically significant change in airway hyperresponsiveness.
  Interventions: Other: ethanol

INTERVENTIONS:
Other: ethanol — subjects will ingest 3 ounces of vodka mixed with fruit juice within 30 min.

SUMMARY:
Alcohol has consequences including increased risk for upper respiratory tract infections, pneumonia, acute respiratory distress syndrome (ARDS), and alcohol-induced asthma. The investigators have established that airways are specifically impacted by alcohol exposure because the airways are heavily exposed to the vapor phase of alcohol during drinking. These preliminary studies demonstrate that brief alcohol administration significantly attenuates airway hyperresponsiveness (AHR) in a mouse model leading to the hypothesis that alcohol exposure modifies airway hyperresponsiveness through a cAMP/NO- dependent mechanism.

DETAILED DESCRIPTION:
Alcohol has well-established consequences in the lung including increased risk for upper respiratory tract infections, pneumonia and acute respiratory distress syndrome (ARDS). There have even been a few reports of alcohol-induced asthma. Data from the investigators' laboratory have established that the airways are specifically impacted by alcohol exposure. Because the airways are heavily exposed to the vapor phase of alcohol during drinking and airway motor tone is modulated by cAMP, the investigators speculated that airway bronchial motor function would be altered in mice fed alcohol. The investigators' preliminary studies demonstrate that brief alcohol administration significantly attenuates airway hyperresponsiveness (AHR) in a mouse model. This novel finding has led us to hypothesize that:

Alcohol exposure modifies airway hyperresponsiveness through a cAMP/NO- dependent mechanism.

ELIGIBILITY:
Inclusion Criteria:

* male
* must be of legal drinking age in the state of Nebraska (≥ 21)
* be between the ages of 21-65
* be non-smokers
* be able to dedicate 3-4 hours on two consecutive days (including waiting at least 2 hours after the alcohol ingestion)
* able to provide informed consent

Exclusion Criteria:

* female
* inability to give informed consent
* any history of lung or allergic disease
* any alcohol intake for the week prior to the experiment
* self-identified history of chronic heavy drinking or alcoholism or psychiatric disorder
* If an otherwise qualifying participant has previously undocumented or unidentified asthma as indicated by the baseline methacholine challenge, that subject will be excluded from the remainder of the study and replaced by another subject

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2013-01-16 (Actual); Study Completion 2013-01-16 (Actual)

PRIMARY OUTCOMES:
Change in airway hyperresponsiveness. | 2 hours
  A one-half concentration difference in the PC20FEV1 will be considered a statistically significant change in airway hyperresponsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Sisson, MD, Study Director — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States